CLINICAL TRIAL: NCT04599218
Title: MR/TRUS Fusion Guided Prostate Biopsy - An Improved Way to Detect and Quantify Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardeshir Rastinehad (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Ardeshir Rastinehad, Associate Professor of Urology and Radiology, Vice Chair of Urology at Lenox Hill Hospital, System Director for Prostate Cancer, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-0384
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Prostate Disease; Elevated Prostate Specific Antigen; Family History of Prostate Cancer; Positive Digital Rectal Exam; Prostate Cancer
Keywords: Prostate Cancer; Prostate Biopsy; Prostate MRI; Targeted Prostate Biopsy; Fusion Biopsy
MeSH Terms: conditions — Prostatic Diseases; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Males with Prostate Cancer (Experimental): Each participant will receive standard of care ultrasound guided prostate biopsy and a MR/TRUS Fusion Guided prostate biopsy.
  Interventions: Other: Prostate Biopsy; Other: MR US Fusion Guided Prostate Biopsy; Device: MR/TRUS Fusion Guided Prostate Biopsy

INTERVENTIONS:
Other: Prostate Biopsy — Standard of care
  Other Names: Transperineal (TP) Prostate Biopsy; UroNav Fusion Biopsy; Targeted prostate biopsy; Ultrasound guided Prostate Biopsy
Other: MR US Fusion Guided Prostate Biopsy — Trans-rectal ultrasound (TRUS) guided fusion prostate biopsy (Arm 1) or a Transperineal Ultrasound guided fusion prostate biopsy (Arm 2). All patients will under go a standard ultrasound guided biopsy at the time of their targeted (fusion) biopsy.
  Other Names: Fusion Biopsy
Device: MR/TRUS Fusion Guided Prostate Biopsy — TRUS images are overlaid on a previously obtained prostate MRI, combined with an electromagnetic tracking system. The urologist then performs directed prostate biopsies at MR-identified targets in addition to the standard prostate biopsies.

SUMMARY:
This research study is designed to determine if targeted Magnetic Resonance Imaging (MRI) Ultrasound (US) fusion biopsy is better than the standard of care ultrasound guided biopsy alone in diagnosing subjects with clinically significant prostate cancer with MRI visible lesions. This study will consist of comparing the standard of care (ultrasound guided prostate biopsy) with the protocol biopsy which consists of an ultrasound guided prostate biopsy and a MRI/US fusion tracked prostate biopsy.

DETAILED DESCRIPTION:
The efficacy of targeting lesions for ultrasound-guided biopsy, surgery,or ablation may be limited by the visibility of a target during the procedure. The successful outcome of the intervention depends upon accurate device placement.

Historically, prostate cancer was diagnosed by finger guided trans-rectal prostate biopsies. However, with the advent of PSA screening and improvements in ultrasonography, ultrasound guided prostate biopsy has become the standard of care to screen and diagnose men with prostate cancer. A standard 12-14 core prostate biopsy is now common practice, detecting cancer in 27% to 44% of patients in patients with an elevated serum PSA.

Initially, prostate MR imaging was not considered for routine clinical practice. However, the addition of an endorectal-coil probe and a 3 Tesla magnet has improved its diagnostic utility. Currently, most mpMRI are done without the use of an endo-rectal coil at 3Tesla. The MRI is able to evaluate the entire prostate (transrectal ultrasound images are overlaid on a previously obtained prostate MRI, combined with an electromagnetic tracking system) prior to biopsy and allows the physician to target specific areas of the prostate that are suspicious for cancer. This contrasts with the typical US guided approach which samples regions of the prostate in a standard fashion.

This study will consist of comparison of the standard of care prostate biopsy with the protocol biopsy which consists of a US guided prostate biopsy and a MR/US fusion tracked prostate biopsy. The researchers are interested in learning which procedure is more useful in obtaining a diagnosis of prostate cancer which will in turn provide a better diagnosis rate. Each patient will act as their own control.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a pre-operative MRI performed in accordance with Northwell/NIH MR Prostate imaging guidelines or equivalent.
2. Age greater than 18 years.
3. No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
4. The ability to understand willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.
5. Ability to tolerate sedation and or general anesthesia if required.
6. PSA >1.8 or Abnormal digital rectal exam or current recommendations or biopsy from the American Urological Association.
7. Pre-Biopsy prostate MRI as described above, showing targetable lesions within 4 months of biopsy
8. Able to tolerate an ultrasound guided biopsy.

Exclusion Criteria:

1. Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study
2. Patients unlikely able to hold reasonably still on a procedure table for the length of the procedure
3. Patients with uncorrectable coagulopathies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1586 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Prostate Cancer | 1 Month
  Incidence of diagnosing subjects with prostate cancer with MR visible lesions

SECONDARY OUTCOMES:
Incidence of adverse events | 1 Month
  the incidence of adverse events occurring after a targeted and ultrasound guided prostate biopsy
Pirads score | 1 Month
  The Prostate Imaging Reporting and Data System (PIRADS) score classifies MRI lesions on a scale from 1 to 5, which reflects their level of suspicion from least to most. Higher score indicates more suspicion.
Gleason score | 1 Month
  The Gleason Score ranges from 1-5 and describes how much the cancer from a biopsy looks like healthy tissue (lower score) or abnormal tissue (higher score). Sum of the gleason grade of the most predominant tumor pattern and a second gleason grade of the second most predominant pattern. Full score from 2 to 10, with higher score indicating more clinically significance.

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Rastinehad, DO, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - The Smith Institute for Urology, Lake Success, New York
  - The Smith Institute for Urology at Lenox Hill, New York, New York
  - Manhattan Eye, Ear, and Throat Hospital (MEETH), New York, New York